CLINICAL TRIAL: NCT04448873
Title: Guided Discontinuation Versus Maintenance Treatment of Sirolimus in Pediatric Patients With Kaposiform Hemangioendothelioma: a Randomized Controlled Trial
Brief Title: Guided Discontinuation Versus Maintenance Treatment of Sirolimus in Pediatric Patients With Kaposiform Hemangioendothelioma
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Children's Hospital of Fudan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LK200421
Record Dates: First submitted 2020-05-10; First posted 2020-06-26 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-09

CONDITIONS: Kaposiform Hemangioendothelioma; Kasabach-Merritt Syndrome
Keywords: Kaposiform Hemangioendothelioma; Kasabach-Merritt Syndrome; Sirolimus; Rapamycin
MeSH Terms: conditions — Kaposiform Hemangioendothelioma; Kasabach-Merritt Syndrome | interventions — Sirolimus

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Only the outcome assessors are blinded, neither clinicians nor patients, because they should be attentive of the risk of relapse in the discontinuation group. Also, it seems unethical if researchers were not to discover the group of patients in the maintenance group who can discontinue sirolimus without relapsing. Clinicians should be given the possibility to adjust dose and ensure the benefits of patients. Therefore, this trial only includes assessors blinding.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Maintenance treatment group (Active Comparator): After at least 2 years of remission of KHE, the participant receives sirolimus as usual. The serum concentration is supposed to be 5-7 ng/ml. If the effect or side effects of sirolimus require discontinuation, it is allowed to modify intervention, and if so, the patient stays in the maintenance group.
  Interventions: Drug: Sirolimus
- Guided discontinuation group (Experimental): After at least 2 years of remission of KHE, the discontinuation measurement should be guided by the clinician with the following principles:
  1. 10% monthly reduction of the previous dose at most.
  2. At least 5 half-lives between each reduction (2 weeks).
  3. Blood concentration should be monitored monthly. Adjustment can be suggested according to the linear relationship between the dose and the blood concentration.
  4. At least 6 months for the duration of guided discontinuation.
  5. Regular assessments and evaluations should be done.
  If the condition relapses or worsens during this process, dose of sirolimus should be adjusted to the previously effective dose. After a 3-month stabilization phase, 5% monthly reduction of the previous dose could be considered.
  Interventions: Drug: Sirolimus

INTERVENTIONS:
Drug: Sirolimus — After at least 2 years of remission of KHE, we compare guided discontinuation with maintenance treatment in pediatric patients with KHE.
  Other Names: Rapamycin

SUMMARY:
This randomized controlled trial aims to compare guided discontinuation with maintenance treatment of sirolimus in pediatric patients with KHE.

DETAILED DESCRIPTION:
Kaposiform Hemangioendothelioma (KHE) is a rare vascular tumor that occurs in infants and children. KHE is characterized by sheets of spindle cells with an infiltrative pattern in the dermis, subcutaneous fat, and muscle. It is locally aggressive and can cause Kasabach-Merritt phenomenon, a serious life-threatening coagulopathy characterized by profound thrombocytopenia and hypofibrinogenemia. Sirolimus, one of the mTOR inhibitors, has become a new and very effective treatment, which is especially reliable for KHE with KMP and has acceptable side effects. However, there is yet no strong evidence on the best practice of treatment length of sirolimus. This randomized controlled trial aims to compare guided discontinuation with maintenance treatment in pediatric patients with KHE in order to provide a basis for the optimal treatment duration of sirolimus, as well as the clinical characteristics of pediatric patients who can safely reduce the dose till withdrawal.

ELIGIBILITY:
Inclusion Criteria:

* Participant diagnosed with KHE with or without KMP
* Participant age 0-12 years
* Participant with detailed medical records of the disease at the time of screening
* Participant with at least two years of remission of KHE and no previous toxicity or adverse events
* Participant with normal liver and kidney function
* Participant with signed and dated informed consent from the guardian(s)

Exclusion Criteria:

* Participant with other hematological diseases
* Participant with other solid tumor
* Participant with general disease such as hypertension, diabetes, adrenal insufficiency, neurological diseases, liver and kidney dysfunction, and cardiopulmonary insufficiency.
* Participant with infectious diseases
* Unwilling participant

Max Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
Remission of KHE and no use of sirolimus at one year follow-up. | From admission to follow-up one year
  The primary outcome is a binary variable. The primary outcome measure will be analyzed with binary logistic regression to estimate the odds ratio between the two groups.

SECONDARY OUTCOMES:
Remission of KHE and the dose of sirolimus at one year follow-up | From admission to follow-up one year
  At one year's follow-up, the participant may be on remission, but still taking sirolimus. The condition is a binary variable and the dose of sirolimus is a continuous variable.
Relapse of KHE and the dose of sirolimus at one year follow-up | From admission to follow-up one year
  At one year's follow-up, the participant may suffer from relapse of KHE and still takes sirolimus. The period of time to the first relapse will be recorded as a time variable, and the cox regression survival analysis model will be used.The dose of sirolimus is a continuous variable. Whether this variable is normally distributed will be checked.
Side effects of sirolimus | From admission to follow-up one year
  The outcome 4 will be described. Adverse events will be reported according to Common Terminology Criteria for Adverse Events, version 4.0 (CTCAE v4.0). Incidence of complications such as oral ulcers, abnormal liver enzymes, infections will be recorded. The blood concentration of sirolimus will be adjusted accordingly.
Platelet count | From admission to follow-up one year
  Platelet count is one of the major indicators of response to treatment and will be used in a prognosis model to predict the clinical characteristics of patients with benefits. It is supposed to be greater than 100×10^9/L.
Fibrinogen level | From admission to follow-up one year
  Fibrinogen level will be used in a prognosis model to predict the clinical characteristics of patients with benefits. It is supposed to be at 2-4g/L.
Tumor volume | From admission to follow-up one year
  Tumor volume will be used in a prognosis model to predict the clinical characteristics of patients with benefits. The size of the tumor is supposed to shrink according to imaging evaluation. The tumor is supposed to be softer by palpation.
Complaints | From admission to follow-up one year
  Complaints are subjective feelings. Whether there is pain, swelling, lameness or skin color change will be recorded as binary variables and used in a prognosis model to predict the clinical characteristics of patients with benefits.

OTHER OUTCOMES:
Remission of KHE and no use of sirolimus at two or three year follow-up | From admission to follow-up two and three years
  This outcome is a binary variable. The primary outcome measure will be analyzed with binary logistic regression to estimate the odds ratio between the two groups.
Remission of KHE and the dose of sirolimus at two or three year follow-up | From admission to follow-up two and three years
  At two or three years' follow-up, the participant may be on remission, but still taking sirolimus. The condition is a binary variable and the dose of sirolimus is a continuous variable.
Relapse of KHE and the dose of sirolimus at two or three year follow-up | From admission to follow-up two and three years
  At two or three years' follow-up, the participant may suffer from relapse of KHE and still takes sirolimus. The period of time to the relapse will be recorded as a time variable, and the cox regression survival analysis model will be used.The dose of sirolimus is a continuous variable. Whether this variable is normally distributed will be checked.

CONTACTS AND LOCATIONS:
Overall Officials: Kai Li, MD, PhD, Principal Investigator — Children's Hospital of Fudan University
Locations (1):
- Children's Hospital of Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wang Z, Yao W, Sun H, Dong K, Ma Y, Chen L, Zheng S, Li K. Sirolimus therapy for kaposiform hemangioendothelioma with long-term follow-up. J Dermatol. 2019 Nov;46(11):956-961. doi: 10.1111/1346-8138.15076. Epub 2019 Sep 5. PMID 31489702
- [Background] Blatt J, Stavas J, Moats-Staats B, Woosley J, Morrell DS. Treatment of childhood kaposiform hemangioendothelioma with sirolimus. Pediatr Blood Cancer. 2010 Dec 15;55(7):1396-8. doi: 10.1002/pbc.22766. PMID 20730884
- [Background] Mauri L, D'Agostino RB Sr. Challenges in the Design and Interpretation of Noninferiority Trials. N Engl J Med. 2017 Oct 5;377(14):1357-1367. doi: 10.1056/NEJMra1510063. No abstract available. PMID 28976859
- [Background] Croteau SE, Liang MG, Kozakewich HP, Alomari AI, Fishman SJ, Mulliken JB, Trenor CC 3rd. Kaposiform hemangioendothelioma: atypical features and risks of Kasabach-Merritt phenomenon in 107 referrals. J Pediatr. 2013 Jan;162(1):142-7. doi: 10.1016/j.jpeds.2012.06.044. Epub 2012 Aug 4. PMID 22871490
- [Background] Schmid I, Klenk AK, Sparber-Sauer M, Koscielniak E, Maxwell R, Haberle B. Kaposiform hemangioendothelioma in children: a benign vascular tumor with multiple treatment options. World J Pediatr. 2018 Aug;14(4):322-329. doi: 10.1007/s12519-018-0171-5. Epub 2018 Jul 27. PMID 30054848
- [Background] Ryu YJ, Choi YH, Cheon JE, Kim WS, Kim IO, Park JE, Kim YJ. Imaging findings of Kaposiform Hemangioendothelioma in children. Eur J Radiol. 2017 Jan;86:198-205. doi: 10.1016/j.ejrad.2016.11.015. Epub 2016 Nov 10. PMID 28027747
- [Background] Ekberg H, Tedesco-Silva H, Demirbas A, Vitko S, Nashan B, Gurkan A, Margreiter R, Hugo C, Grinyo JM, Frei U, Vanrenterghem Y, Daloze P, Halloran PF; ELITE-Symphony Study. Reduced exposure to calcineurin inhibitors in renal transplantation. N Engl J Med. 2007 Dec 20;357(25):2562-75. doi: 10.1056/NEJMoa067411. PMID 18094377
- [Background] Gianfreda D, Nicastro M, Galetti M, Alberici F, Corradi D, Becchi G, Baldari G, De Filippo M, Ferretti S, Moroni G, Foti R, Di Gangi M, Jeannin G, Saffroy R, Emile JF, Buzio C, Vaglio A. Sirolimus plus prednisone for Erdheim-Chester disease: an open-label trial. Blood. 2015 Sep 3;126(10):1163-71. doi: 10.1182/blood-2015-01-620377. Epub 2015 Jun 3. PMID 26041743
- [Background] Brahmer JR, Lacchetti C, Schneider BJ, Atkins MB, Brassil KJ, Caterino JM, Chau I, Ernstoff MS, Gardner JM, Ginex P, Hallmeyer S, Holter Chakrabarty J, Leighl NB, Mammen JS, McDermott DF, Naing A, Nastoupil LJ, Phillips T, Porter LD, Puzanov I, Reichner CA, Santomasso BD, Seigel C, Spira A, Suarez-Almazor ME, Wang Y, Weber JS, Wolchok JD, Thompson JA; National Comprehensive Cancer Network. Management of Immune-Related Adverse Events in Patients Treated With Immune Checkpoint Inhibitor Therapy: American Society of Clinical Oncology Clinical Practice Guideline. J Clin Oncol. 2018 Jun 10;36(17):1714-1768. doi: 10.1200/JCO.2017.77.6385. Epub 2018 Feb 14. PMID 29442540
- [Background] Sturup AE, Jensen HD, Dolmer S, Birk M, Albert N, Nielsen M, Hjorthoj C, Eplov L, Ebdrup BH, Mors O, Nordentoft M. TAILOR - tapered discontinuation versus maintenance therapy of antipsychotic medication in patients with newly diagnosed schizophrenia or persistent delusional disorder in remission of psychotic symptoms: study protocol for a randomized clinical trial. Trials. 2017 Sep 29;18(1):445. doi: 10.1186/s13063-017-2172-4. PMID 28962668
- [Background] Wang D, Chen X, Li Z. Population pharmacokinetics of sirolimus in pediatric patients with kaposiform hemangioendothelioma: A retrospective study. Oncol Lett. 2019 Sep;18(3):2412-2419. doi: 10.3892/ol.2019.10562. Epub 2019 Jul 4. PMID 31452734
- [Background] MacDonald A, Scarola J, Burke JT, Zimmerman JJ. Clinical pharmacokinetics and therapeutic drug monitoring of sirolimus. Clin Ther. 2000;22 Suppl B:B101-121. doi: 10.1016/s0149-2918(00)89027-x. PMID 10823378
- [Background] Holt DW, Mandelbrot DA, Tortorici MA, Korth-Bradley JM, Sierka D, Levy DI, See Tai S, Horowitz GL. Long-term evaluation of analytical methods used in sirolimus therapeutic drug monitoring. Clin Transplant. 2014 Feb;28(2):243-51. doi: 10.1111/ctr.12305. Epub 2014 Jan 30. PMID 24476346
- [Background] Mariani LG, Schmitt IR, Garcia CD, Kiszewski AE. Low dose sirolimus treatment for refractory tufted angioma and congenital kaposiform hemangioendothelioma, both with Kasabach-Merritt phenomenon. Pediatr Blood Cancer. 2019 Aug;66(8):e27810. doi: 10.1002/pbc.27810. Epub 2019 May 14. No abstract available. PMID 31087627
- [Background] Mizuno T, Emoto C, Fukuda T, Hammill AM, Adams DM, Vinks AA. Model-based precision dosing of sirolimus in pediatric patients with vascular anomalies. Eur J Pharm Sci. 2017 Nov 15;109S:S124-S131. doi: 10.1016/j.ejps.2017.05.037. Epub 2017 May 17. PMID 28526601